CLINICAL TRIAL: NCT01451268
Title: Phase I/II Study With Oral Panobinostat Maintenance Therapy Following Allogeneic Stem Cell Transplantation in Patients With High Risk MDS or AML (PANOBEST)
Brief Title: Phase I/II Study With Oral Panobinostat Maintenance Therapy Following Allogeneic Stem Cell Transplantation in Patients With High Risk Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML)
Acronym: PANOBEST
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Gesine Bug, Senior physician hematology, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589 BDE05T
Record Dates: First submitted 2011-09-30; First posted 2011-10-13 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: 60 to 150 Days After Allogeneic Stem Cell Transplantation; High Risk MDS; MDS; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panobinostat Arm A (Experimental)
  Interventions: Drug: Panobinostat
- Panobinostat Arm B (Experimental)
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — 10mg upto 40mg Panobinostat dose escalation in consequent cohorts; frequency: three times a week, every week; duration: one year
  Other Names: LBH589
  Arms: Panobinostat Arm A
Drug: Panobinostat — Start of Arm B after completion of Arm A; initial dose-level: one level below MTD of Arm A; 10mg upto 60mg Panobinostat dose escalation in consequent cohorts; frequency: three times a week, every other week; duration: one year
  Other Names: LBH589
  Arms: Panobinostat Arm B

SUMMARY:
The study's primary objective is to determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of Panobinostat when administered within 150 days after hematopoietic stem cell transplantation (HSCT) and given in conjunction with standard immunosuppressive therapy after HSCT for patients with high-risk Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML).

Secondary objectives are

* To determine safety and tolerability of panobinostat
* To determine overall and disease-free survival at 12 months after HSCT
* To evaluate immunoregulatory properties of panobinostat
* To evaluate patient-reported health-related quality of life (HRQL)

The hypothesis of this study is that panobinostat can be an effective drug in preventing relapse of MDS and AML patients with high-risk features after hematopoietic stem cell transplantation with reduced-intensity conditioning (RIC-HSCT) while at the same time reducing graft-versus-host disease (GvHD) with preservation of graft-versus-leukemia (GvL) effect.

ELIGIBILITY:
Inclusion Criteria:

* AML (except acute promyelocytic leukemia, AML M3) with high-risk features defined as one or more of the following criteria:

  * refractory to or relapsed after at least one cycle of standard chemotherapy
  * > 10% bone marrow blasts at day 15 of the first induction cycle
  * adverse risk cytogenetics including complex karyotype (≥ 3 abnormalities or abnormalities of chromosomes 3, 5 or 7) regardless of stage
  * secondary to MDS or radio-/chemotherapy or
* MDS RAEB according to the WHO classification or intermediate-2 or high-risk according to IPSS or
* Chronic myelomonocytic leukemia (CMML) with ≥ 5% bone marrow blasts and

  * Allogeneic HSCT with reduced intensity conditioning (see Section 15.1 for definition) performed within 60 - 150 days prior to study entry
  * Complete hematologic remission documented by bone marrow aspiration within 28 days prior to study entry

Exclusion Criteria:

* Active acute GvHD overall grade 2 - 4
* Prior treatment with a deacetylase (DAC) inhibitor
* Patients with impaired cardiac function or other concurrent severe and/or uncontrolled medical conditions
* Clinical symptoms suggesting central nervous system (CNS) leukemia
* Patient has an impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of panobinostat | after 28 days of administration
Dose-limiting toxicity (MTD) of Panobinostat | after 28 days of administration

SECONDARY OUTCOMES:
Cumulative incidence of hematologic relapse and death | one year after HSCT
Reconstitution of the immune system as measured by changes in numbers, ratio, phenotype and activation state of peripheral blood cell populations during panobinostat therapy | patients will be followed for up to 2 years depending on the duration of study participation
Time to complete donor chimerism | patients will be followed for up to 2 years depending on the duration of study participation
Cumulative incidence of extensive chronic GvHD | one year after HSCT
Duration of complete donor chimerism | patients will be followed for up to 2 years depending on the duration of study participation
Cumulative incidence of severe acute GvHD | one year after HSCT
patient-reported health-related quality of life | after 3 months of administration and one month after last intake of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Gesine Bug, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (6):
- Germany (6):
  - University Hospital Düsseldorf, Düsseldorf
  - University Hospital Essen, Essen
  - University Hospital Frankfurt, Frankfurt am Main
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital Mainz, Mainz
  - University Hospital Marburg, Marburg

REFERENCES:
- See also: Trial register of the Kompetenznetz Leukämien, additional trial information — http://www.studienregister-online.de